CLINICAL TRIAL: NCT05362734
Title: Freeze All Strategy Versus Fresh Embryo Transfer After GnRH Analogue Trigger
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 999
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Hyperstimulation Syndrome; Pregnancy Related
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First fresh embryo transfer (group A): The two groups analysed were defined according to the modality of first embryo transfer: cycles in which a fresh ET was performed at first, after a dual triggering or a rescue protocol (Group A) and cycles where a frozen-thawed ET was performed at first, after being chosen a freeze-all strategy (Group B).
  Interventions: Behavioral: obstetric outcomes after fresh versus cryopreserved embryo transfer
- First cryopreserved embryo transfer (group B): The two groups analysed were defined according to the modality of first embryo transfer: cycles in which a fresh ET was performed at first, after a dual triggering or a rescue protocol (Group A) and cycles where a frozen-thawed ET was performed at first, after being chosen a freeze-all strategy (Group B).
  Interventions: Behavioral: obstetric outcomes after fresh versus cryopreserved embryo transfer

INTERVENTIONS:
Behavioral: obstetric outcomes after fresh versus cryopreserved embryo transfer — measure of ongoing pregnancy rate, delivery rate, abortion rate, ectopic pregnancy rate, multiple birth rate, ovarian hyperstimulation syndrome incidence, drop out rate

SUMMARY:
Ovarian hyperstimulation syndrome (OHSS) is one of the most dangerous complications of assisted reproduction technology (ART), described in approximatively 3 to 10% of stimulation cycles although an underestimation of the real incidence has been suggested.

The use in clinical practice of GnRH antagonist has made it possible to perform the trigger with GnRH analogues, with the advantage of considerably reducing the risk of OHSS.

DETAILED DESCRIPTION:
The main concerns about the trigger with analogue are about obstetric outcomes, since it may increase the Abortion Rate (AR) and reduce the Ongoing Pregnancy Rate (OPR) due to luteal phase deficiency, and on the other hand about oocyte quality and competence.

While in order to maximize the chance of pregnancy at fresh embryo transfer after GnRHa trigger, several studies have focused on the importance of luteal phase support, other authors suggest that the best strategy is freeze-all: cryopreservation of all the obtained embryos and subsequent single embryo transfers.

However, data about oocyte quality, retrieval rate, pregnancy rate and reduced occurrence of complications such as OHSS, especially on the very first embryo transfer, are still scarce.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ART cycle with antagonist protocol stimulation and trigger with GnRH agonist
* patients are believed at risk of OHSS at time of trigger based on size and number of follicles developed (≥18 follicles with diameter 12 mm at induction).

Exclusion Criteria:

* hypogonadotropic hypogonadism
* other ART protocols
* any patient that underwent freeze-all strategy in order to perform pre-implantation genetic testing (PGT)
* oncological or deferring motherhood freezing procedures

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study database includes all Oocyte Retrievals (OR) performed between 01/01/2012 and 31/12/2020 at Humanitas Fertility Center after antagonist protocol stimulation and trigger with GnRH agonist.
Sampling Method: Non-Probability Sample
Enrollment: 1396 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 8 years
  number of viable pregnancies that had completed at least 12 weeks of gestation on the total number of ETs performed
delivery rate | 8 years
  number of deliveries of one or more live births over the total performed ET

SECONDARY OUTCOMES:
Other pregnancy outcomes | 8 years
  ectopic pregnancy rate, miscarriage rate, multiple Birth Rate
Safety profile | 8 years
  Severe ovarian hyperstimulation syndrome incidence
the dropout rate | 8 years
  number of cycles in which any live birth (from either ART and/or spontaneous conceive) was not achieved and still some embryos or oocytes had to be thawed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kupka MS, Ferraretti AP, de Mouzon J, Erb K, D'Hooghe T, Castilla JA, Calhaz-Jorge C, De Geyter C, Goossens V; European IVF-Monitoring Consortium, for the European Society of Human Reproduction and Embryology. Assisted reproductive technology in Europe, 2010: results generated from European registers by ESHREdagger. Hum Reprod. 2014 Oct 10;29(10):2099-113. doi: 10.1093/humrep/deu175. Epub 2014 Jul 27. PMID 25069504
- [Background] Humaidan P, Nelson SM, Devroey P, Coddington CC, Schwartz LB, Gordon K, Frattarelli JL, Tarlatzis BC, Fatemi HM, Lutjen P, Stegmann BJ. Ovarian hyperstimulation syndrome: review and new classification criteria for reporting in clinical trials. Hum Reprod. 2016 Sep;31(9):1997-2004. doi: 10.1093/humrep/dew149. Epub 2016 Jun 23. PMID 27343272
- [Background] Levi-Setti PE, Di Segni N, Gargasole C, Ronchetti C, Cirillo F. Ovarian Hyperstimulation: Diagnosis, Prevention, and Management. Semin Reprod Med. 2021 Nov;39(5-06):170-179. doi: 10.1055/s-0041-1736492. Epub 2021 Oct 13. PMID 34644798
- [Background] De Geyter C, Calhaz-Jorge C, Kupka MS, Wyns C, Mocanu E, Motrenko T, Scaravelli G, Smeenk J, Vidakovic S, Goossens V; European IVF-monitoring Consortium (EIM) for the European Society of Human Reproduction and Embryology (ESHRE). ART in Europe, 2015: results generated from European registries by ESHRE. Hum Reprod Open. 2020 Feb 24;2020(1):hoz038. doi: 10.1093/hropen/hoz038. eCollection 2020. PMID 32123753
- [Background] Humaidan P, Kol S, Papanikolaou EG; Copenhagen GnRH Agonist Triggering Workshop Group. GnRH agonist for triggering of final oocyte maturation: time for a change of practice? Hum Reprod Update. 2011 Jul-Aug;17(4):510-24. doi: 10.1093/humupd/dmr008. Epub 2011 Mar 30. PMID 21450755
- [Background] Humaidan P, Bredkjaer HE, Bungum L, Bungum M, Grondahl ML, Westergaard L, Andersen CY. GnRH agonist (buserelin) or hCG for ovulation induction in GnRH antagonist IVF/ICSI cycles: a prospective randomized study. Hum Reprod. 2005 May;20(5):1213-20. doi: 10.1093/humrep/deh765. Epub 2005 Mar 10. PMID 15760966
- [Background] Lawrenz B, Coughlan C, Fatemi HM. Individualized luteal phase support. Curr Opin Obstet Gynecol. 2019 Jun;31(3):177-182. doi: 10.1097/GCO.0000000000000530. PMID 30855289
- [Background] Abbara A, Islam R, Clarke SA, Jeffers L, Christopoulos G, Comninos AN, Salim R, Lavery SA, Vuong TNL, Humaidan P, Kelsey TW, Trew GH, Dhillo WS. Clinical parameters of ovarian hyperstimulation syndrome following different hormonal triggers of oocyte maturation in IVF treatment. Clin Endocrinol (Oxf). 2018 Jun;88(6):920-927. doi: 10.1111/cen.13569. Epub 2018 Mar 6. PMID 29446481
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517
- [Background] ESHRE Special Interest Group of Embryology and Alpha Scientists in Reproductive Medicine. Electronic address: coticchio.biogenesi@grupposandonato.it. The Vienna consensus: report of an expert meeting on the development of ART laboratory performance indicators. Reprod Biomed Online. 2017 Nov;35(5):494-510. doi: 10.1016/j.rbmo.2017.06.015. Epub 2017 Aug 4. PMID 28784335
- [Background] ESHRE Clinic PI Working Group; Vlaisavljevic V, Apter S, Capalbo A, D'Angelo A, Gianaroli L, Griesinger G, Kolibianakis EM, Lainas G, Mardesic T, Motrenko T, Pelkonen S, Romualdi D, Vermeulen N, Tilleman K. The Maribor consensus: report of an expert meeting on the development of performance indicators for clinical practice in ART. Hum Reprod Open. 2021 Jul 3;2021(3):hoab022. doi: 10.1093/hropen/hoab022. eCollection 2021. PMID 34250273
- [Background] Tomas C, Alsbjerg B, Martikainen H, Humaidan P. Pregnancy loss after frozen-embryo transfer--a comparison of three protocols. Fertil Steril. 2012 Nov;98(5):1165-9. doi: 10.1016/j.fertnstert.2012.07.1058. Epub 2012 Jul 27. PMID 22840239
- [Background] ESHRE working group on Ectopic Pregnancy; Kirk E, Ankum P, Jakab A, Le Clef N, Ludwin A, Small R, Tellum T, Toyli M, Van den Bosch T, Jurkovic D. Terminology for describing normally sited and ectopic pregnancies on ultrasound: ESHRE recommendations for good practice. Hum Reprod Open. 2020 Dec 16;2020(4):hoaa055. doi: 10.1093/hropen/hoaa055. eCollection 2020. PMID 33354626
- [Background] Committee on Practice Bulletins-Gynecology. ACOG Practice Bulletin No. 191: Tubal Ectopic Pregnancy. Obstet Gynecol. 2018 Feb;131(2):e65-e77. doi: 10.1097/AOG.0000000000002464. PMID 29232273
- [Background] Sunkara SK, Zheng W, D'Hooghe T, Longobardi S, Boivin J. Time as an outcome measure in fertility-related clinical studies: long-awaited. Hum Reprod. 2020 Aug 1;35(8):1732-1739. doi: 10.1093/humrep/deaa138. PMID 32644107